CLINICAL TRIAL: NCT05467423
Title: Single Center Clinical Trial to Evaluate the Effect of Low-dose Versus Standard-dose Iron Supplementation on the Gut Microbiome in Non-anemic Iron-deficient Females
Brief Title: Effect of Low-dose Versus Standard-dose Iron Supplementation on the Gut Microbiome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Pierre-Alexandre Krayenbuehl, Professor Pierre-Alexandra Krayenbuehl, University of Zurich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IronGutMicrobiome
Record Dates: First submitted 2022-07-05; First posted 2022-07-20 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Iron Deficiency (Without Anemia)
Keywords: Iron; Microbiome; Gut Bacteria
MeSH Terms: conditions — Iron Deficiencies | interventions — Iron

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard-dose (Active Comparator): The standard-dose arm takes one 100mg of iron per day together with a meal, no matter breakfast, lunch or dinner - one tablet a day.
  Interventions: Dietary Supplement: Iron
- Low-dose (Experimental): The low-dose arm 12mg of iron a day. The first 6mg tablet in the morning on an empty stomach and the second 6mg tablet in the evening either one hour before or after eating - two tablets a day.
  Interventions: Dietary Supplement: Iron

INTERVENTIONS:
Dietary Supplement: Iron — 4 weeks of daily oral iron therapy. The subjects administer the therapy themselves.

SUMMARY:
Iron deficiency is a common problem that is often treated with the administration of oral iron.

Most of the iron is not absorbed and remains in the intestine, where it influences the balance of gut bacteria.

This influence is usually undesirable and should be kept as small as possible. With lower iron doses, the amount of unabsorbed iron is smaller and therefore a smaller change in the intestinal bacteria composition is to be expected.

DETAILED DESCRIPTION:
Iron deficiency affects about one in five premenopausal women. The first line treatment for patients with iron deficiency is an oral therapy with iron-supplements, another option is the intravenous iron supplementation.

The oral supplementation causes side-effects such as nausea, vomiting, abdominal pain and many more in a lot of patients. There is a positive correlation between the appearance of gastrointestinal side-effects and the applicated iron dose.

Only a low fraction of orally taken iron is actually absorbed, even in patients with iron-deficiency. Since only a fraction of the orally administered iron is actually absorbed, the toxicity of high concentrations of iron in the gastrointestinal tract and the altered selection advantages of the bacteria presumably leads to microbiome changes.

The unabsorbed iron is potentially changing the microbiome, which leads to undesirable side effects.

With low-dose iron-supplementation the amount of unabsorbed iron is smaller, therefore a dosage dependent microbiome change would be expected.

The aim of the study is to determine the magnitude of the microbiome response to daily iron substitution with 12mg and 100mg.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Female gender
* Premenopausal
* Age > 18 years
* Regular menstrual cycle
* BMI in normal range (18-25kg/m2)
* Serum-ferritin ≤30ng/ml
* No anemia (hemoglobin ≥117g/l)
* No intake of dietary supplements for at least 4 weeks

Exclusion Criteria:

* Pregnancy
* Hypermenorrhea (more than 5 unties/tampons per day)
* Chronic inflammatory disease, psychiatric disorders
* Hypersensitivity to iron supplements
* chronic kidney disease (creatinine >80 µmol/l)
* Liver disease (ALT >35 U/l)
* Hypo- or Hyperthyroidism (TSH not between 0.16-4.25 mU/l)
* Intake of medicines that interact with oral iron supplementation (e.g. PPI)*

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-01-04 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Microbiome diversity and oral iron therapy | 4 weeks
  The microbiome is analyzed using stool samples. A stool sample is taken before and after the 4 weeks period. The low-dose arm is expected to have a smaller decrease compared to the standard-dose arm. The microbiome composition is measured using 16S rDNA gene amplicon sequencing. The results are analysed using the Shannon-Index to include diversity as well as abundance.

SECONDARY OUTCOMES:
Side-effects of treatment | 4 weeks
  Adverse events will be assessed on a report form after 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsspital Zürich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No